CLINICAL TRIAL: NCT03956069
Title: Study of the Diagnostic Value of "Rapid" High Throughput Genome Sequencing Analysis in Diagnostic Emergency Situations
Acronym: FASTGEN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: SORLIN PHRCI 2018
Record Dates: First submitted 2019-05-15; First posted 2019-05-20 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Developmental Anomalies
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: blood sample — for patient and its parents
Genetic: genome sequencing — whole genome sequencing

SUMMARY:
Rare diseases (affecting less than one in 2,000 people) are a major public health issue. There are about 8,000 rare diseases and they affect more than 3 million people in France. Most of these diseases are diagnosed in children, and they are responsible for 10% of deaths before the age of 5. Up to 80% of these diseases are believed to be of genetic origin. New generation high throughput sequencing (HTS) technologies, which allow the study of an individual's entire genome, have emerged in recent years as a tool of choice for the study of rare diseases. Our team was the first in France to demonstrate the value of exome sequencing (ES: all coding regions (exons), representing 1% of the total genome size) in the diagnosis of severe diseases in pediatric patients, developmental anomalies and intellectual disability.

Although it represents a significant advance in the diagnosis of genetic diseases, ES provides a contributing result in only about 30% of cases in patients with no obvious clinical diagnosis and with normal CGH-array. Sequencing the entire genome (GS) promises to improve the ability to study the causes of genetic diseases, with an expected diagnostic rate of 50 to 60% through the concomitant identification of point variations, CNVs and structural variations. While some international teams have already implemented GS in the diagnosis of rare diseases, only two teams report the use of trio GS in emergency situations in the neonatal period, with a low yield for first-line diagnostic use (31 and 42% respectively). It is therefore essential that these preliminary results be compared with other studies before considering the deployment of GS in diagnostic, early detection or rapidly evolving emergency situations, such as neonatal resuscitation or pediatric neurological distress.

ELIGIBILITY:
Inclusion Criteria:

* Children (0-6 years old) hospitalized in neonatal intensive care or pediatric intensive care with a suspected genetic disease and without an obvious clinical diagnosis
* Possibility of taking the proband and their 2 biological parents
* Parents affiliated to or beneficiaries of the national health insurance system
* Informed consent signed by the legal representatives of the minor patient
* Ability to understand the study for both biological parents

Exclusion Criteria:

* Diagnostic hypothesis considered highly probable with an available molecular test having a lower cost than GS
* Individuals who have already had high throughput sequencing (panel, ES)
* Parents protected
* Families where one of the two holders of parental authority is not a biological parent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: child with a suspected genetic disease without an obvious clinical diagnosis and both biological parents
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
identification of a causal diagnosis | Through study completion, an average of 2 years
  identification of genetic etiology

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France